CLINICAL TRIAL: NCT04425616
Title: SafeFit Trial: Virtual Clinics to Deliver Universal Interventions to Maintain and Improve Mental and Physical Health in People With Cancer Who Are Following Social Distancing Guidance: A COVID-19 Targeted Trial
Brief Title: SafeFit Trial: Virtual Clinics to Deliver Universal Interventions in People With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Macmillan Cancer Support (Other); CanRehab Trust (Unknown); Wessex Cancer Alliance (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RHM CRI 0403
Record Dates: First submitted 2020-06-03; First posted 2020-06-11 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2023-11

CONDITIONS: Cancer; COVID
Keywords: COVID-19; Virtual clinics; Exercise; Cancer diagnosis; Nutrition; Psychological support; Behaviour change
MeSH Terms: conditions — Neoplasms; COVID-19; Motor Activity | interventions — Exercise; Nutritional Status

STUDY DESIGN:
Intervention Model Description: Non-randomised phase III interventional trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Universal Interventions (Experimental): The delivery of nutrition, exercise and psychological interventions delivered in the following structure:
  * Month 1: Up to three times per week
  * Months 2-3: Once per week
  * Months 4 - 6: One session per month for the last 3 months
  Interventions: Other: Exercise; Behavioral: Psychological and Behaviour Change Support; Other: Nutrition

INTERVENTIONS:
Other: Exercise — At least one and up to three supervised sessions per week including:
  * aerobic exercise at a rating of perceived exertion of 11-14 (6-20 scale) accumulating 20 minutes per session
  * resistance exercise of 8-10 exercises for 2x 8-15 repetitions performed in a controlled manner and covering the whole body
  * Range of motion exercise performed through pain free range of motion covering the whole body to be maintained in good alignment for 10-30 seconds, with some movements held for a second set of 10-30 seconds if stiff
Behavioral: Psychological and Behaviour Change Support — Instructors will be trained in Healthy Conversation Skills (HCS), Making Every Contact Count (MECC) or equivalent. This will enable them to deliver brief participant centred empowering interventions informed by social cognitive theory. This skill set will be used to support participants in adopting and maintaining the prescribed exercise and diet programme as well as adopting and practicing strategies to self-manage psychological well-being. Participants will be given the option to be provided with a SMARTER goal setting sheet to assist with goal planning. Applicable standardised psychological support resources will be made available to the participants though the Macmillan resource repository that they can access online or in alternative format as necessary, for example relaxation and mindfulness exercises
Other: Nutrition — Instructors will receive training in generic nutritional principles in line with recommendations from World Cancer Research Fund (WCRF) and British Dietetic Association, and will work with participant to review own diet and eating habits against WCRF recommendations to enable goal setting and identify links to existing resources reputable websites, outputs and on-line forums. These would include: principles of healthy eating ('eat well' advice), weight management, symptom management, prehab advice before treatment starts, rehab advice during and after treatment. The participant will be asked if they are eating and drinking well or have any concerns at the beginning of each exercise session. Further support will be provided to instructors to address participant concerns or requests for additional information.

SUMMARY:
Trial Phase: Phase III: Interventional Trial: Virtual clinics to deliver universal interventions to maintain and improve physical health, nutritional state and psychological wellbeing in people with cancer who are following social distancing guidance: A COVID-19 targeted trial.

Indication: Male or female participants, aged over 18 years old with suspicion or confirmed diagnosis of cancer (does not require histological confirmation)

Objective: To investigate the efficacy of remote multimodal universal interventions delivered via virtual clinics to improve physical function as measured by the EORTC-QLQ-C30.

Secondary Objective:

To investigate the efficacy of remote multimodal universal interventions delivered via virtual clinics to improve emotional function, quality of life, participant activation (PAM), behaviour change and the effect it has on health economics (EQ-5D-5L).

Exploratory Objective:

Overall Survival and adherence to the intervention/advice using validated tools or development of a web-based toolkit.

DETAILED DESCRIPTION:
Rationale: A recent statement by Professor Chris Whitty, Chief Medical Officer, NHS England, emphasised the significant benefits of exercise for all people. He said, "this may be challenging for people self-isolating and even more so for those highly vulnerable people that are having to shield against the virus in their own homes" The coronavirus (COVID-19) pandemic has led to many changes to everyday life including the introduction of social distancing as well as restriction of travel. Treatment plans for patients with cancer are being revised or modified due to risks and benefits of certain treatments in light of the COVID-19 risk. The number of deaths due to the disruption in cancer services is likely to outweigh the number of deaths from coronavirus itself over the next five years.

The effects of this pandemic has reportedly led to increased anxiety and distress and risks deconditioning due to reduced physical activity. The interventions we are proposing aim to enable people with cancer to optimise their physical health, nutritional state and psychological wellbeing and prepare for their treatment pathway (current or modified) and recovery during this uncertain time through exercise, nutrition and psychological support.

The aim is to investigate whether the promotion of these interventions delivered via virtual clinics, in socially distanced people with cancer, can improve physical and psychological function and self-efficacy to self-manage. We are also aiming to evaluate health economics whilst following the COVID-19 government guidelines.

Trial Design: Phase III: Non randomised Interventional Trial

Sample Size: 1100

Intervention: Provision of dietary, exercise and psychological advice as well as behaviour change support (universal interventions) as aligned to the universal interventions (with the caveats of COVID-19) in the Macmillan 'Principles and guidance for prehabilitation within the management and support of people with cancer' guideline. This complex intervention will be prescribed and delivered through virtual clinics where CanRehab professionals will support the individual. Level 3 Personal Trainers may also deliver the interventions in some cases with a GP referral qualification and who are competent in delivering the interventions to participants with cancer post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, aged over 18 years old
* Suspicion or confirmed diagnosis of cancer (does not require histological confirmation)

Exclusion Criteria:

- Participants unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Physical Function | Baseline up to 1 year post enrolment
  Physical function will be measured using the EORTC-QLQ-C30. Participants will choose from the choices 1 = Not at all; 2 = A little, 3 = Quite a bit, 4 = Very much

SECONDARY OUTCOMES:
Emotional Function | Baseline up to 1 year post enrolment
  Emotional function will be measured using the EORTC-QLQ-C30. Participants will choose from the choices 1 = Not at all; 2 = A little, 3 = Quite a bit, 4 = Very much
Health related quality of life | Baseline up to 1 year post enrolment
  EQ-5D-5L is a standardised measure of health status developed by the EuroQol Group. Applicable to a wide range of health conditions and treatments, it provides a simple descriptive profile and a single index value for health status that can be used in the clinical evaluation of health care
Health economics analysis | Baseline up to 1 year post enrolment
  EQ-5D-5L is a standardised measure of health status developed by the EuroQol Group. Applicable to a wide range of health conditions and treatments, it provides a simple descriptive profile and a single index value for health status that can be used in the economic evaluation of health care
Patient activation | Baseline up to 1 year post enrolment
  Patients knowledge skills and confidence to manage their own health and care will be measured using the Patient Activation Measure (PAM)
  Agreement or disagreement with statements. Choice between disagree strongly, disagree, agree, agree strongly and not applicable
Self-reported physical activity | Baseline up to 1 year post enrolment
  Measured using the Godin Leisure Time Exercise Questionnaire, a 7-day physical activity recall
Nutrition assessment | Baseline up to 1 year post enrolment
  In the oncology population where malnutrition prevalence is high, the Patient-Generated Subjective Global Assessment Short Form (PG-SGA SF) is a descriptive screening tool that can provide further information to assist triaging and capture acute change in nutritional state
Self-efficacy for self-management of chronic disease | Baseline up to 1 year post enrolment
  Self-efficacy (confidence) to self-manage chronic disease (SEMCD), measured using the Lorig SEMCD scale
  A confidence scale that represents the patients confidence that a regular task can be achieved. 1 = Not confident at all and 10= totally confident.
Distress levels | Baseline up to 1 year post enrolment
  Levels of distress as measured by the Emotions Thermometers. Participants will score on a scale where 0 = None and 10 = Extreme
Functional capacity | Baseline up to 1 year post enrolment
  The Dukes Activity Status Index is a 12 item self-report measure of functional capacity that can be used to estimate peak oxygen uptake
The impact of COVID-19 pandemic on psychological functioning | Baseline up to 1 year post enrolment
  As measured by the Impact of Event Scale - a 22-item self-report measure of the imapact of a specific traumatic event against the DSM criteria for Post Traumatic Stress Disorder. 0 = Not at all and 4 = Extremely.
Process Evaluation | Through study completion, an average of 12 months
  Semi-structured interviews with participants and professionals to explore acceptability, usefulness and barriers to delivery/engagement

OTHER OUTCOMES:
Exploratory: Overall survival | 1 year post enrolment
  Overall survival at 1 year following date of enrolment
Exploratory: Adherence to the interventions/advice | Baseline up to 1 year post enrolment
  Adherence to intervention advice is defined as number of sessions the participants attends divided by the total number of sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Southampton NHS FT, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grimmett C, Bates A, West M, Leggett S, Varkonyi-Sepp J, Campbell A, Davis J, Wootton S, Shaw C, Barlow R, Ashcroft J, Scott A, Moyes H, Hawkins L, Levett DZH, Williams F, Grocott MPW, Jack S. SafeFit Trial: virtual clinics to deliver a multimodal intervention to improve psychological and physical well-being in people with cancer. Protocol of a COVID-19 targeted non-randomised phase III trial. BMJ Open. 2021 Aug 26;11(8):e048175. doi: 10.1136/bmjopen-2020-048175. PMID 34446487